CLINICAL TRIAL: NCT01676441
Title: A Phase II/III Clinical Trial to Evaluate the Safety and Efficacy of Bone Marrow-derived Mesenchymal Stem Cell Transplantation in Patients With Chronic Spinal Cord Injury.
Brief Title: Safety and Efficacy of Autologous Mesenchymal Stem Cells in Chronic Spinal Cord Injury
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: sponsor decision (confidential)
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cerecellgram-spine
Record Dates: First submitted 2012-08-23; First posted 2012-08-31 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; mesenchymal stem cell
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: posterior cervical laminectomy and Mesenchymal stem cells(cellgram-spine) tranplantation.
  After laminectomy, 1.6X107 and 3.2 X107 Autologous Mesenchymal stem cells is injected into the intramedullary and intrathecal space respectively
Oversight: Data Monitoring Committee: No

ARMS (1):
- cellgram-spine (Experimental): posterior cervical laminectomy and Mesenchymal stem cells tranplantation. After laminectomy, 1.6X10^7 and 3.2 X10^7 Autologous Mesenchymal stem cells is injected into the intramedullary and intrathecal space respectively
  Interventions: Drug: cellgram-spine

INTERVENTIONS:
Drug: cellgram-spine — Mesenchymal stem cells transplantation
  Other Names: Mesenchymal stem cells

SUMMARY:
This phase II/III clinical trial is designed to evaluate the safety and efficacy of autologous Mesenchymal Stem Cells (MSC) transplanted directly into the injured spinal cord.

DETAILED DESCRIPTION:
The Principal investigator has performed a clinical trial using autologous MSCs in patients with cervical spinal cord injury. The results revealed the safety of autologous MSC. This Phase II, III single-center trial is to assess the safety and efficacy of bone marrow-derived mesenchymal stem cell transplantation direct to injured spinal cord site via laminectomy. After recovery from the operation, the subjects receive 4 weeks of physical and occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 16-65 years
* Traumatic spinal cord injury at the level of cervical
* American Spinal Injury Association Impairment Scale B
* 12 months or more post spinal cord injury subject with stable neurological finding after more than 1 month rehabilitation therapy
* No signs of contracture
* Good physical condition to go through operation
* Must be willing and able to participate in study procedures with no mental and verbal problem
* Able to consent by patients or legal representatives

Exclusion Criteria:

* Serum SGOT/SGPT > 3 X upper limit of normal or Creatinine > 1.5 X upper limit of normal
* Major surgical procedure in the past 3 months
* Penetrating injury
* Mechanical ventilation
* Serious pre-existing medical conditions
* Recently diagnosed infection (Urinary tract infection, Pneumonia etc)
* Positive skin test for penicillin
* Positive result for viral markers (human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and Venereal Disease Research Laboratory (VDRL) test)
* Pregnant women, women of childbearing potential who do not want adequate contraception, breastfeeding females
* Unwilling to participate in study
* Patients with psychiatric disorder severe as to make compliance with the treatment unlike, and signing informed consent impossible
* Drug abuse in the past 1 year
* Participating in other clinical trials in the past 1 month
* Inappropriate patients to participate in the study according to the chief investigator

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Compared change of Motor Score of the American Spinal Injury Association (ASIA) scale | Baseline, post operation(24 hours), 1 month, 3 month, 6 month, 12 month
  Compared Baseline and after 6, 12 months of cell treatment, ASIA motor test analyzes the proportion of patients with a motor grade of more than 2 devision, with a motor grade improving from 2 to 3 and a rise of 5 or more in total score.
  <American Spinal Injury Association (ASIA) scale> 0 Total paralysis
  1. Palpable or visible contraction
  2. Active movement, full Range Of Motion(ROM) with gravity eliminated
  3. Active movement, full ROM against gravity
  4. Active movement, full ROM against gravity and moderate resistance in a muscle specific position
  5. (normal) Active movement, full ROM against gravity and full resistance in a functional muscle position expected from an otherwise unimpaired person 5* (normal) Active movement, full ROM against gravity and sufficient resistance to be considered normal if identified inhibiting factors (i.e. pain, disuse) were not present NT Not testable

SECONDARY OUTCOMES:
Sensory score of the American Spinal Injury Association (ASIA) scale | Baseline, post operation(24 hours), 1 month, 3 month, 6 month, 12 month
  Analyze the difference between the pre and post of the ASIA sensory score by using the Study's pre-test (Wilcoxon's signed test).
  <American Spinal Injury Association (ASIA) scale> The exam is based on neurological responses, touch and pinprick sensations tested in each dermatome, and strength of the muscles that control key motions on both sides of the body. Sensation is graded on a scale of 0-2: 0 is no sensation, 1 is altered or decreased sensation, and 2 is full sensation. Each side of the body is graded independently. When an area is not available (e.g. because of an amputation or cast), it is recorded as "NT", "not testable".
Electrophysiological change (Motor Evoked Potentials-MEP, Somatosensory Evoked Potentials-SSEP) | 6 months
  Post 6 months of treatment, the validity is analyzed through patients who have expressed their responses to the electrophysiological test (Motor Evoked Potentials-MEP, Somatosensory Evoked Potentials-SSEP).
MRI and Diffusion Tensor Imaging of spinal cord | 6 months
  Post 6 months of cell treatment, the ratio of patients with changes in magnetic resonance imaging is analyzed.

OTHER OUTCOMES:
Number of adverse events | Baseline to 12 months
  Analyze the laboratory, vital sign, ECG, physical exam, medical exam, chest X-ray results from baseline to end of the study for investigate adverse reactions and view safety.

CONTACTS AND LOCATIONS:
Overall Officials: Sangryong Jeon, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

REFERENCES:
- [Background] Park JH, Kim DY, Sung IY, Choi GH, Jeon MH, Kim KK, Jeon SR. Long-term results of spinal cord injury therapy using mesenchymal stem cells derived from bone marrow in humans. Neurosurgery. 2012 May;70(5):1238-47; discussion 1247. doi: 10.1227/NEU.0b013e31824387f9. PMID 22127044